CLINICAL TRIAL: NCT02707991
Title: Nurse Case Management to Improve Linkage to Hepatitis C Care and Treatment Initiation in HIV Co-infection: A Randomized Controlled Trial
Brief Title: Nurse Case Management to Improve Hepatitis C Care in HIV Co-infection
Acronym: Care2Cure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IRB00081068
Record Dates: First submitted 2016-03-09; First posted 2016-03-15 (Estimated); Results first posted 2019-05-02 (Actual); Last update posted 2019-05-02 (Actual); Status verified 2019-01

CONDITIONS: HIV; Hepatitis C, Chronic
Keywords: Continuity of Patient Care; Treatment Cascade
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Usual Care (No Intervention): Usual clinic appointment process plus receipt of the Centers for Disease Control and Prevention (CDC) Hepatitis C Fact Sheet
- Nurse Case Management (Experimental): Nurse-initiated hepatitis C clinic referral, strengths-based education, patient navigation, appointment reminders, and care coordination of HIV/hepatitis C drug-drug interaction prevention
  Interventions: Behavioral: Nurse Case Management

INTERVENTIONS:
Behavioral: Nurse Case Management — Participants will receive one baseline nurse case management study visit in addition to appointment reminders one week and one day before the scheduled hepatitis clinic appointment. Those who link to the Viral Hepatitis Clinic and are identified as eligible to start hepatitis C therapy by their health care provider will have one additional study visit with the nurse case manager to coordinate drug-drug interaction prevention.
  Other Names: Care Coordination
  Arms: Nurse Case Management

SUMMARY:
Effective all-oral medications are finally available to cure hepatitis C virus, which affects more than 4 million Americans and one-in-four people living with HIV. However, many barriers exist that prevent people with HIV/HCV co-infection from getting this curative treatment, including low knowledge, competing demands, and drug interactions with HIV medications.

This study evaluates if a hepatitis C nurse case management intervention in an HIV primary care clinic will improve patient attendance to hepatitis C care and help people start hepatitis C treatment earlier. Half of the participants will receive brief case management with a nurse, while the other half will receive usual clinic care.

DETAILED DESCRIPTION:
Hepatitis C virus (HCV) is a leading cause of liver cancer and HCV-related liver disease is among the most common causes of non-AIDS related death among people living with HIV (PLWH). One quarter of PLWH in the U.S. are co-infected with HCV, which leads to a 3-fold increase in progression to end stage liver disease and liver cancer. HCV can be cured, but less than half of PLWH with chronic HCV in the U.S. have linked to HCV care, and about 7% initiated treatment. Poor treatment initiation rates historically have been due to low efficacy among PLWH, but HCV care now is at a turning point. The investigators have the ability to substantially decrease HCV-related morbidity and mortality in PLWH with the availability of effective all-oral treatment. As patients are funneled into HCV care, improving the process of linkage to care and treatment preparation related to HIV medication modifications necessary for current HCV regimens is essential to maximize the lifesaving potential of available therapies among PLWH.

There are several barriers to linkage to HCV care and treatment. HCV is a "silent epidemic" often presenting no symptoms for 20 years. Knowledge about HCV and its available therapies is also low and lags behind new advancements in HCV treatment. Competing work, school and caregiving demands has also historically led to low motivation to engage in HCV care. For PLWH who are linked to HCV care, drug interactions between new HCV therapies and HIV treatment regimens introduce a new barrier to HCV treatment initiation. Up to 88% of PLWH will need to switch their HIV treatment regimen to avoid contraindicated drug interactions. The April 8, 2015 Guidelines for the Use of Antiretroviral Agents in HIV-1-infected Adults and Adolescents emphasize the need to modify HIV regimens to treat HCV in many PLWH. But modifying HIV treatment regimens can have severe negative consequences, including decreased quality of life, increased symptom burden, and loss of viral suppression.

Interventions that both increase HCV knowledge and support HIV treatment modifications in the setting of drug interactions are needed to improve linkage to HCV care and decrease time to treatment initiation. In similar settings and populations, nurse case management interventions have been shown to improve these outcomes. However, few of these interventions have been rigorously tested in the context of HCV.

This study is a randomized, single-blinded controlled trial to test whether a nurse case management intervention will improve the HCV treatment cascade among PLWH in an HIV primary care setting compared to usual care.

Specifically, this study aims to:

1. Test whether a nurse case management intervention will increase linkage to the Viral Hepatitis Clinic among persons with HIV/HCV co-infection compared to usual care; Hypothesis: A higher proportion of those who are randomized to the intervention arm will attend the Viral Hepatitis Clinic within 60 days of randomization compared to those who receive usual care.
2. Determine if a nurse case management intervention will decrease time to HCV treatment initiation among persons with HIV/HCV co-infection compared to usual care; Hypothesis: Those who are randomized to the intervention arm will have a decreased time to HCV treatment initiation from the point of randomization compared to those who receive usual care.
3. Describe the characteristics associated with uptake of HCV care among people living with HIV, controlling for covariates; Research question 2.1: What patient-level characteristics are associated with increased uptake of HCV care?; Research question 2.2: Compared to the known historical barriers to engaging in HCV care, what factors continue to be associated with uptake of HCV care in the new paradigm of HCV treatment for people living with HIV?

ELIGIBILITY:
Inclusion Criteria:

* HIV infection
* Chronic hepatitis C infection
* Did not attend a hepatitis C specialty appointment in the past year
* Able to speak English
* Current patient at the John G. Bartlett Specialty Practice at Johns Hopkins Hospital (at least 1 visit in the past year)

Exclusion Criteria:

* Pregnancy
* Emergency medical care needed
* Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason E Farley, PhD, MPH, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yehia BR, Schranz AJ, Umscheid CA, Lo Re V 3rd. The treatment cascade for chronic hepatitis C virus infection in the United States: a systematic review and meta-analysis. PLoS One. 2014 Jul 2;9(7):e101554. doi: 10.1371/journal.pone.0101554. eCollection 2014. PMID 24988388
- [Background] Patel N, Nasiri M, Koroglu A, Amin R, McGuey L, McNutt LA, Roman M, Miller C. Prevalence of drug-drug interactions upon addition of simeprevir- or sofosbuvir-containing treatment to medication profiles of patients with HIV and hepatitis C coinfection. AIDS Res Hum Retroviruses. 2015 Feb;31(2):189-97. doi: 10.1089/AID.2014.0215. Epub 2015 Jan 6. PMID 25432275
- [Background] Cachay ER, Hill L, Ballard C, Colwell B, Torriani F, Wyles D, Mathews WC. Increasing Hepatitis C treatment uptake among HIV-infected patients using an HIV primary care model. AIDS Res Ther. 2013 Mar 28;10(1):9. doi: 10.1186/1742-6405-10-9. PMID 23537147
- [Background] Ly KN, Xing J, Klevens RM, Jiles RB, Ward JW, Holmberg SD. The increasing burden of mortality from viral hepatitis in the United States between 1999 and 2007. Ann Intern Med. 2012 Feb 21;156(4):271-8. doi: 10.7326/0003-4819-156-4-201202210-00004. PMID 22351712
- [Background] Lo Re V 3rd, Kallan MJ, Tate JP, Localio AR, Lim JK, Goetz MB, Klein MB, Rimland D, Rodriguez-Barradas MC, Butt AA, Gibert CL, Brown ST, Park L, Dubrow R, Reddy KR, Kostman JR, Strom BL, Justice AC. Hepatic decompensation in antiretroviral-treated patients co-infected with HIV and hepatitis C virus compared with hepatitis C virus-monoinfected patients: a cohort study. Ann Intern Med. 2014 Mar 18;160(6):369-79. doi: 10.7326/M13-1829. PMID 24723077
- [Background] Thomas DL. Cure of hepatitis C virus infection without interferon alfa: scientific basis and current clinical evidence. Top Antivir Med. 2014 Jan;21(5):152-6. PMID 24531555
- [Background] Mehta SH, Genberg BL, Astemborski J, Kavasery R, Kirk GD, Vlahov D, Strathdee SA, Thomas DL. Limited uptake of hepatitis C treatment among injection drug users. J Community Health. 2008 Jun;33(3):126-33. doi: 10.1007/s10900-007-9083-3. PMID 18165889
- [Background] Afdhal NH, Zeuzem S, Schooley RT, Thomas DL, Ward JW, Litwin AH, Razavi H, Castera L, Poynard T, Muir A, Mehta SH, Dee L, Graham C, Church DR, Talal AH, Sulkowski MS, Jacobson IM; New Paradigm of HCV Therapy Meeting Participants. The new paradigm of hepatitis C therapy: integration of oral therapies into best practices. J Viral Hepat. 2013 Nov;20(11):745-60. doi: 10.1111/jvh.12173. PMID 24168254
- [Background] Harris M, Rhodes T. Hepatitis C treatment access and uptake for people who inject drugs: a review mapping the role of social factors. Harm Reduct J. 2013 May 7;10:7. doi: 10.1186/1477-7517-10-7. PMID 23651646
- [Background] Swan D, Long J, Carr O, Flanagan J, Irish H, Keating S, Keaveney M, Lambert J, McCormick PA, McKiernan S, Moloney J, Perry N, Cullen W. Barriers to and facilitators of hepatitis C testing, management, and treatment among current and former injecting drug users: a qualitative exploration. AIDS Patient Care STDS. 2010 Dec;24(12):753-62. doi: 10.1089/apc.2010.0142. PMID 21138381
- [Background] Munoz-Plaza CE, Strauss S, Astone-Twerell J, Jarlais DD, Gwadz M, Hagan H, Osborne A, Rosenblum A. Exploring drug users' attitudes and decisions regarding hepatitis C (HCV) treatment in the U.S. Int J Drug Policy. 2008 Feb;19(1):71-8. doi: 10.1016/j.drugpo.2007.02.003. Epub 2007 Aug 6. PMID 18312822
- [Background] Fusfeld L, Aggarwal J, Dougher C, Vera-Llonch M, Bubb S, Donepudi M, Goss TF. Assessment of motivating factors associated with the initiation and completion of treatment for chronic hepatitis C virus (HCV) infection. BMC Infect Dis. 2013 May 23;13:234. doi: 10.1186/1471-2334-13-234. PMID 23701894
- [Background] Wagner G, Osilla KC, Garnett J, Ghosh-Dastidar B, Bhatti L, Witt M, Goetz MB. Provider and patient correlates of provider decisions to recommend HCV treatment to HIV co-infected patients. J Int Assoc Physicians AIDS Care (Chic). 2012 Jul-Aug;11(4):245-51. doi: 10.1177/1545109712444163. Epub 2012 May 7. PMID 22564797
- [Background] Rockstroh JK. Optimal therapy of HIV/HCV co-infected patients with direct acting antivirals. Liver Int. 2015 Jan;35 Suppl 1:51-5. doi: 10.1111/liv.12721. PMID 25529087
- [Background] Chen EY, North CS, Fatunde O, Bernstein I, Salari S, Day B, Jain MK. Knowledge and attitudes about hepatitis C virus (HCV) infection and its treatment in HCV mono-infected and HCV/HIV co-infected adults. J Viral Hepat. 2013 Oct;20(10):708-14. doi: 10.1111/jvh.12095. Epub 2013 Apr 1. PMID 24010645
- [Background] Craw JA, Gardner LI, Marks G, Rapp RC, Bosshart J, Duffus WA, Rossman A, Coughlin SL, Gruber D, Safford LA, Overton J, Schmitt K. Brief strengths-based case management promotes entry into HIV medical care: results of the antiretroviral treatment access study-II. J Acquir Immune Defic Syndr. 2008 Apr 15;47(5):597-606. doi: 10.1097/QAI.0b013e3181684c51. PMID 18285714
- [Background] Gardner LI, Metsch LR, Anderson-Mahoney P, Loughlin AM, del Rio C, Strathdee S, Sansom SL, Siegal HA, Greenberg AE, Holmberg SD; Antiretroviral Treatment and Access Study Study Group. Efficacy of a brief case management intervention to link recently diagnosed HIV-infected persons to care. AIDS. 2005 Mar 4;19(4):423-31. doi: 10.1097/01.aids.0000161772.51900.eb. PMID 15750396
- [Background] Tyler D, Nyamathi A, Stein JA, Koniak-Griffin D, Hodge F, Gelberg L. Increasing hepatitis C knowledge among homeless adults: results of a community-based, interdisciplinary intervention. J Behav Health Serv Res. 2014 Jan;41(1):37-49. doi: 10.1007/s11414-013-9333-3. PMID 23616250
- [Background] Gupta K, Romney D, Briggs M, Benker K. Effects of a brief educational program on knowledge and willingness to accept treatment among patients with hepatitis C at inner-city hospitals. J Community Health. 2007 Aug;32(4):221-30. doi: 10.1007/s10900-007-9046-8. PMID 17696047
- [Background] Holtzman CW, Shea JA, Glanz K, Jacobs LM, Gross R, Hines J, Mounzer K, Samuel R, Metlay JP, Yehia BR. Mapping patient-identified barriers and facilitators to retention in HIV care and antiretroviral therapy adherence to Andersen's Behavioral Model. AIDS Care. 2015;27(7):817-28. doi: 10.1080/09540121.2015.1009362. Epub 2015 Feb 11. PMID 25671515
- [Background] Finitsis DJ, Pellowski JA, Johnson BT. Text message intervention designs to promote adherence to antiretroviral therapy (ART): a meta-analysis of randomized controlled trials. PLoS One. 2014 Feb 5;9(2):e88166. doi: 10.1371/journal.pone.0088166. eCollection 2014. PMID 24505411
- [Background] Andersen RM. Revisiting the behavioral model and access to medical care: does it matter? J Health Soc Behav. 1995 Mar;36(1):1-10. PMID 7738325
- [Background] Masson CL, Delucchi KL, McKnight C, Hettema J, Khalili M, Min A, Jordan AE, Pepper N, Hall J, Hengl NS, Young C, Shopshire MS, Manuel JK, Coffin L, Hammer H, Shapiro B, Seewald RM, Bodenheimer HC Jr, Sorensen JL, Des Jarlais DC, Perlman DC. A randomized trial of a hepatitis care coordination model in methadone maintenance treatment. Am J Public Health. 2013 Oct;103(10):e81-8. doi: 10.2105/AJPH.2013.301458. Epub 2013 Aug 15. PMID 23947319
- [Background] Gottlieb LN. Strengths-based nursing. Am J Nurs. 2014 Aug;114(8):24-32; quiz 33,46. doi: 10.1097/01.NAJ.0000453039.70629.e2. PMID 25036663
- [Background] Farley JE, Kelly AM, Reiser K, Brown M, Kub J, Davis JG, Walshe L, Van der Walt M. Development and evaluation of a pilot nurse case management model to address multidrug-resistant tuberculosis (MDR-TB) and HIV in South Africa. PLoS One. 2014 Nov 18;9(11):e111702. doi: 10.1371/journal.pone.0111702. eCollection 2014. PMID 25405988
- See also: AASLD/IDSA Recommendations for Testing, Managing, and Treating Hepatitis C — http://hcvguidelines.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place from July 2016 to February 2018 in an outpatient infectious disease clinic in Baltimore, Maryland
Period: Overall Study
Arm/Group | Enhanced Usual Care | Nurse Case Management
Started | 33 | 35
Day 60 Data Collectio | 32 | 34
Month 6 Data Collection | 32 | 34
Completed | 32 | 34
Not Completed | 1 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Became ineligible | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Enhanced Usual Care | Nurse Case Management | Total
Number analyzed (Participants) | 33 | 35 | 68
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 33 | 63
  >=65 years | 3 | 2 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.32 (7.73) | 54.76 (7.68) | 55.03 (7.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 26
  Male | 20 | 22 | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 31 | 35 | 66
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 26 | 29 | 55
  White | 4 | 6 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 33 | 35 | 68
HIV viral load [Count of Participants; unit: Participants] — HIV plasma ribonucleic acid (RNA) not detectable (less than 20 copies/milliliter)
  Participants | 15 | 14 | 29
Liver fibrosis level [Count of Participants; unit: Participants] — The fibrosis score is used to describe the amount of inflammation in the liver. A lower score (F0) is more desirable than a higher score (F4):
  F0: No fibrosis F1: Portal fibrosis without septa F2: Portal fibrosis with few septa F3: Numerous septa without cirrhosis F4: Cirrhosis
  Participants
    Less than F2 | 7 | 7 | 14
    Greater than or equal to F2 | 13 | 11 | 24
    Unknown | 13 | 17 | 30
Health insurance [Count of Participants; unit: Participants] — Currently enrolled in Medicaid and/or Medicare
  Participants | 33 | 34 | 67
Hepatitis C knowledge [Mean (Standard Deviation); unit: units on a scale] — Total score on the Brief Hepatitis C Knowledge Scale: A point is given for each correct answer on this true/false scale, with a maximum possible number of points (perfect score) of 19 and a minimum number of points (no questions answered correctly) of 0.
  units on a scale | 15.39 (2.01) | 14.83 (2.12) | 15.10 (2.07)
Alcohol use [Count of Participants; unit: Participants] — Self-reported drinking alcohol in the past 12 months
  Participants | 10 | 18 | 28
Injection drug use [Count of Participants; unit: Participants] — Self-reported using drugs intravenously in the past 12 months
  Participants | 9 | 7 | 16

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Linked to Care
Description: This will be assessed based on the number of participants who attend an appointment at the Viral Hepatitis Clinic within 60 days of enrolling in the study. A participant is considered "linked to care" if he/she attends an appointment at the clinic. A participant is considered "not linked to care" if he/she does not attend an appointment at the clinic. Whether a participant linked to care will be determined by looking at the medical record, where all attended appointments are documented. If no attended appointment is documented, this will be considered non-attendance/not linked to care.
Time Frame: 60 days
Population: All eligible participants who were randomized are included. Two participants were excluded (one in each arm) because they were found to be ineligible for study participation after they were randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced Usual Care | Nurse Case Management
Number analyzed (Participants) | 32 | 34
Participants | 8 | 16
Statistical Analysis 1: Comparison: Enhanced Usual Care vs Nurse Case Management; Test type: Superiority; p = 0.036, z-test for difference in proportions — one-sided test; Mean Difference (Final Values) = 22, Standard Error of Mean 0.115

2. Secondary Outcome: Time to Hepatitis C Treatment Initiation
Description: Number of days from study enrollment to receipt of the first dose of hepatitis C treatment
Time Frame: 6 months
Population: ll eligible participants who were randomized are included. Two participants were excluded (one in each arm) because they were found to be ineligible for study participation after they were randomized.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Enhanced Usual Care | Nurse Case Management
Number analyzed (Participants) | 32 | 34
days | 103 (48.5) | 79.3 (26.8)

ADVERSE EVENTS:
Time Frame: 6 months
Description: Data were collected via a monthly medical record review
Arm/Group | Enhanced Usual Care | Nurse Case Management
All-Cause Mortality (participants affected / at risk) | 0/33 | 2/35
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/35
Other Adverse Events (participants affected / at risk) | 0/33 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-08): https://cdn.clinicaltrials.gov/large-docs/91/NCT02707991/Prot_SAP_000.pdf